CLINICAL TRIAL: NCT05778877
Title: Phase 1/2 Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of SEL-302 (MMA-101 Following Administration of SEL-110) in Pediatric Subjects With Mut Subtype Isolated Methylmalonic Acidemia (MMA)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of SEL-302 in Pediatric Subjects With MMA
Acronym: reiMMAgine
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decided by sponsor
Sponsor: Selecta Biosciences, Inc. (Industry)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SEL-302.101; 000957-HG (Other: NHGRI)
Record Dates: First submitted 2023-01-23; First posted 2023-03-21 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Methylmalonic Acidemia (MMA)
Keywords: MMA; gene therapy; methylmalonic acidemia; adeno associated virus; organic acidemia; Methylmalonyl-CoA Mutase
MeSH Terms: conditions — Methylmalonic acidemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Adolescents (Experimental): IV infusion of MMA-101 in the first patient on Day 1 IV infusion of SEL-302 in the second and third patient on Day 1, followed by two repeat doses of SEL-110 on Day 28 and Day 56 Adolescents ages ≥12 and <18
  Interventions: Drug: SEL-302
- Cohort 2 - Children (Experimental): IV infusion of SEL-302 in all patients on Day 1, followed by two repeat doses of SEL-110 on Day 28 and Day 56 Children ages ≥3 and <12
  Interventions: Drug: SEL-302

INTERVENTIONS:
Drug: SEL-302 — SEL-302 Drug: MMA-101 (1.0E13 vg/kg)
  Drug: SEL-110 (0.15 mg/kg or up to 0.3 mg/kg)
  Other Names:
  SEL-110.36, ImmTOR
  Other Names: AAV8-MMUT

SUMMARY:
This Phase 1/2 study will evaluate the safety and pharmacodynamics (PD) of SEL-302, which consists of the gene transfer vector MMA-101 following administration of an immunomodulatory SEL-110 agent in pediatric subjects with Methylmalonyl-CoA Mutase (MMUT) MMA.

DETAILED DESCRIPTION:
MMA is a rare inborn error of branched chain amino acid metabolism. Despite strict dietary adherence and vigilant monitoring and care, affected individuals have recurrent episodes of severe illness and develop complications from different organ systems that can be life-threatening. Liver transplants can help, but gene transfer therapy could offer an alternative treatment option. This study will be an open-label, single dose, single center study of SEL-302 consisting of two investigative therapeutics: a gene transfer therapy that is using an inactive virus, called adeno-associated-virus 8 (AAV8), to deliver the MMUT gene to the liver, by itself called MMA-101, and an immunotherapy called SEL-110, a nano-encapsulated form of sirolimus.

The study will enroll two cohorts treating up to a total of 6 subjects.

Cohort 1: 3 adolescents (≥12 and <18 years of age) Cohort 2: 3 children (≥3 and <12 years of age, with a minimum body weight of 15 kg)

The dose of MMA-101 administered to each subject will be 1.0E13 vg/kg. Each progression to the next subject dosed in the study will be reviewed and approved by a data safety monitoring committee.

The first subject in Cohort 1 will receive only MMA-101. The second adolescent subject in Cohort 1 will be treated with 0.15 mg/kg of SEL-110 followed by MMA-101 on Day 1 and two repeat doses of 0.15 mg/kg of SEL-110 at Day 28 and Day 56. The dose of SEL-110 in the third subject in Cohort 1 may be increased up to 0.3 mg/kg depending on results from the second subject. After assessment of safety and efficacy of Cohort 1, Cohort 2 will be started in younger children.

The dose of SEL-110 in Cohort 2 for the first subject will be 0.15 mg/kg of SEL-110 immediately prior to the dose of MMA-101 on Day 1 and two repeat doses of 0.15 mg/kg of SEL-110 at Day 28 and Day 56. The dose of SEL-110 in the second and third subject in Cohort 2 may be increased up to 0.3 mg/kg at one or more of the three doses depending on results of all previously treated subjects.

The primary efficacy endpoints of reduction in serum methylmalonic acid (sMMA) levels and increases in the 1-13C sodium propionate oxidation breath test (POBT) will be assessed at an interim timepoint for safety evaluation (Day 84) and at the primary endpoint of 1 year.

All subjects will be monitored closely for safety for the first year of the study and then annually for an additional 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to <18 years at time of consent (assent where possible)
2. Confirmed diagnosis of MMUT type methylmalonic acidemia by molecular genetic testing
3. Clinical and biochemical diagnosis of severe MMA as defined by:

   1. sMMA level between 100 to 3,000 μmol/L
   2. A clinical history consistent with severe MMA
   3. Subjects must have fully recovered from any hospitalization for metabolic ketoacidosis or surgery at least 4 weeks prior to the start of the screening period.
   4. Parent or legal guardian are willing and able to provide informed consent. Written assent will be obtained from minors older than age seven whenever possible.
   5. Subject and caregiver must be willing to comply with study-related assessments and adhere to lifestyle considerations throughout study duration.

Exclusion Criteria:

1. History of any organ transplantation.
2. High MMUT liver enzymatic activity in the range seen in healthy subjects or MMA patients after corrective liver transplant, as demonstrated by POBT levels.
3. Presence of Nab against AAV8 or polyethylene glycol (PEG)
4. An estimated glomerular filtration rate (GFR)<45 mL/min/1.73 m2 (<chronic kidney disease stage 3a)
5. Hemoglobin <10 g/dL
6. Platelet count <100,000 per mm3
7. History of any malignancy or immunocompromising condition.
8. History of anaphylaxis or severe allergic reaction to drug therapy, foods, PEG or polysorbates.
9. Previously received gene therapy or messenger ribonucleic acid (mRNA) treatments for MMA.
10. Participated in a clinical trial of another (non-gene or mRNA therapy) investigational agent within 30 days prior to screening, or within 5 elimination half-lives of the investigational agent, whichever is longer.

Note: additional inclusion/exclusion criteria may apply, per protocol.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SEL-302 | From the initial administration of SEL-302 up to 5 years for long-term follow-up.
  Incidence and severity of all adverse events (AEs), treatment emergent AEs (TEAEs), and serious adverse events (SAEs) and their relationship to SEL-302 (MMA-101 or SEL-110) Time Frame: From the initial administration of SEL-302 up to 5 years for long-term follow-up.
PD Activity of SEL-302 | From initial treatment with SEL-302 up to 5 years for long-term follow-up.
  Measure the change in sMMA levels at Day 84 (interim endpoint for safety assessment) and at the end of the 1-year study period (primary endpoint) and assessed yearly during the 4 years of long-term follow-up.
PD Activity of SEL-302 | From initial treatment with SEL-302 up to 5 years for long-term follow-up.
  Measure the change in the 1-13C sodium POBT at Day 84 (interim endpoint for safety assessment) and at the end of the 1-year study period (primary endpoint) and assessed yearly during the 4 years of long-term follow-up.
Assess the change in Neutralizing antibody (Nab) titers for MMA-101 with treatment of SEL-110 | From initial treatment with SEL-302 up to 5 years for long-term follow-up.
  Measure Nab serum titers from baseline at multiple timepoints following treatment on Day 28, Day 56, and Day 84.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of sirolimus | From initial treatment with SEL-302 up to 84 days following administration of SEL-110.
  Measuring the Cmax of sirolimus at the first, second, and third dose of SEL-110.
  Time Frame: From initial treatment with SEL-302 up to 84 days following administration of SEL-110.
Area Under Curve (AUC) of sirolimus | From initial treatment with SEL-302 up to 84 days following administration of SEL-110.
  Measuring the AUC of sirolimus at the first, second, and third dose of SEL-110.
Patient outcomes assessed by the frequency and severity of specified clinical events | From initial treatment with SEL-302 up to 5 years for long-term follow-up.
  Recording of patient outcomes regarding metabolic crisis in need of sick-day dietary modifications, hospitalization, and need for referral for liver, kidney, or liver/kidney transplant.
World Health Organization Quality of Life Brief Version (WHOQoL-BREF) | From initial treatment with SEL-302 for up to 5 years for long-term follow-up.
  Assess the change from baseline in patient-reported quality of life measures using the WHOQoL-BREF (on a number scale of 0 to 100, with lower indicating a worse outcome).
Zarit Burden Interview | From initial treatment with SEL-302 for up to 5 years for long-term follow-up.
  Assess the change from baseline in patient-reported quality of life measures using the Zarit Burden Interview (on a number scale from 0 to 48, with higher indicating a greater burden)

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute, National Institutes of Health, Bethesda, Maryland, United States